CLINICAL TRIAL: NCT01192009
Title: Leucine and Skeletal Muscle Disuse: Clinical Anti-Atrophic Effectiveness and Related Mechanisms
Brief Title: Leucine Supplementation and Skeletal Muscle Disuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Humberto Nicastro, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009/02896-6
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Disuse Atrophy
Keywords: Leucine; Skeletal Muscle Disuse; Atrophy; Proteolysis
MeSH Terms: conditions — Muscular Disorders, Atrophic; Atrophy | interventions — Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immobilization and Leucine (Experimental)
  Interventions: Dietary Supplement: Leucine
- Immobilization and Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Leucine — 7.2 g of leucine during 2 weeks
  Arms: Immobilization and Leucine
Dietary Supplement: Placebo — 7.2 g of alanine during 2 weeks
  Arms: Immobilization and Placebo

SUMMARY:
Leucine supplementation is widely known for promoting strong influence on skeletal muscle remodeling. This study aims to evaluate the effect of leucine supplementation on disuse-induced skeletal muscle atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of anterior cruciate ligament injury
* Physically active
* Must be able to swallow tablets
* Non-smokers
* Do not use nutritional supplements

Exclusion Criteria:

* Post-surgical complications

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle structure (cross-sectional area) | 2 weeks

SECONDARY OUTCOMES:
Molecular signalling pathways (hypertrophy, atrophy, and inflammation) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Humberto Nicastro, PhD Student, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo - School of Physical Education and Sports, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Zanchi NE, Nicastro H, Lancha AH Jr. Potential antiproteolytic effects of L-leucine: observations of in vitro and in vivo studies. Nutr Metab (Lond). 2008 Jul 17;5:20. doi: 10.1186/1743-7075-5-20. PMID 18637185
- [Background] Nicastro H, Artioli GG, Costa Ados S, Solis MY, da Luz CR, Blachier F, Lancha AH Jr. An overview of the therapeutic effects of leucine supplementation on skeletal muscle under atrophic conditions. Amino Acids. 2011 Feb;40(2):287-300. doi: 10.1007/s00726-010-0636-x. Epub 2010 Jun 1. PMID 20514547